CLINICAL TRIAL: NCT05281146
Title: Production of Fortified Biscuit With Chickpea and Crushed Peanut and Evaluating Its Effectiveness in Terms of Its Acceptability and Cognitive Performance: a Pilot Study Among Egyptian Primary School-aged Children
Brief Title: Production of Fortified Biscuit With Chickpea and Crushed Peanut for Improving Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Prof.Dr. Ammal Mokhtar Metwally, Prof. Public Health and Community Medicine, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180926
Record Dates: First submitted 2022-02-28; First posted 2022-03-16 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Performance
Keywords: chickpea; crushed peanut; Wheat germ; Cinnamon; short-term memory; working memory; visual memory; information processing; auditory attention ability

STUDY DESIGN:
Intervention Model Description: Theoretically, fortified biscuits based on chickpea flour and crushed peanuts in addition to wheat germ, and Cinnamon help in enhancing immunity, fighting viruses, maintaining regular and healthy bowel movement, regulating blood sugar and cholesterol levels, and more importantly improving cognitive abilities of school aged children. It is important to practically evaluate the effectiveness of the fortified biscuits intake for 4 months in terms of its acceptability and impact on cognitive performance for a sample of children aged 8-12 years attending rural primary schools in an Egyptian village. Eighty Children were randomly allocated in either chickpea and peanuts biscuits dependent group (40 children) or the non-dependent group (40 children).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chickpea and peanuts biscuits dependent group (Active Comparator): children aged 8- 12 years attending the village school. This group received one daily pack of three fortified biscuits as snakes between breakfast and lunch on daily basis for four months.
  Interventions: Dietary Supplement: Chickpeas and crushed peanuts fortified biscuit; Other: Cognitive stimulation for the mothers; Other: Cognitive stimulation for students
- The chickpea and crushed peanut biscuits non-dependent group (Active Comparator): Matched age and sex children attending the same village school. This group did not receive the fortified biscuits but received their ordinary usual breakfasts or snacks for four months.
  Interventions: Other: Cognitive stimulation for the mothers; Other: Cognitive stimulation for students

INTERVENTIONS:
Dietary Supplement: Chickpeas and crushed peanuts fortified biscuit — This group received one daily pack of three fortified biscuits as snakes between breakfast and lunch on daily basis for four months. The chickpeas and crushed peanuts fortified biscuit consisted of wheat flour (extract 72%), Chickpea flour, crushed peanuts, wheat germ, Skimmed milk, corn oil, egg, sugar, Cinnamon, baking powder, salt, and vanilla.
  Arms: chickpea and peanuts biscuits dependent group
Other: Cognitive stimulation for the mothers — I. Sessions for mothers
  * Informing mothers about the most common causes of poor school achievement
  * Clarification of mother's and family roles in improving student's cognitive abilities
  * Defining cognitive functions needed for learning and school achievement
    o Attention, perceptive reasoning, memory, problem solving, proper use of language
  * Identifying sensory functions necessary for the growth of cognitive functions
  * Explaining factors that assist in academic excellence
Other: Cognitive stimulation for students — * Activities to improve focus and visual attention
  * Activities to improve visual memory
  * Activities to improve vigilance and auditory attention
  * Explaining types of memory Causes of weak memory Factors helping in improving memory Nutritional elements improving memory
  * Training on skills of problem-solving

SUMMARY:
It is well known that globally, school-based fortification and school feeding approaches have been applied to remedy nutritional deficiencies that impact health in the primary school age group.

Aim of the study: to produce a fortified biscuit with chickpea and crushed peanut. To evaluate the effectiveness of the fortified biscuits intake for 4 months in terms of its acceptability and impact on cognitive performance for a sample of children aged 8-12 years attending rural primary schools in an Egyptian village. The fortified biscuits' effect on auditory attention, visual and working memory, and learning ability was evaluated.

Methodology: This study was an interventional study conducted in two stages: stage one was the production of nutritious biscuits that is based on chickpea flour and peanut in addition to whole wheat (extract 72 %), wheat germ, cinnamon, milk, and egg. All these constituents help in enhancing immunity, fighting viruses, maintaining regular and healthy bowel movement, regulating blood sugar and cholesterol levels, and more importantly improving the cognitive abilities of school-aged children. During stage two, eighty Children were randomly allocated in either chickpea and peanuts biscuits dependent group (40 children) or non-dependent group (40 children) to evaluate the impact of the fortified biscuits. All enrolled children and their mothers received 5 cognitive stimulation sessions over four months. The cognitive performance of primary school-aged children was assessed before and after the interventions by a battery of four verbal & non-verbal intelligence psychological tests. These tests covered short-term and working memory, visual memory, and the ability for categorization, learning for speed of information processing, and auditory attention ability with rising levels of difficulty. These tests were: Digit Span, the figural memory tests, Coding and Auditory vigilance tests A and B respectively. Five items were used to evaluate the physical characteristics of the biscuits: color, odor, taste, consistency, and general acceptance.

DETAILED DESCRIPTION:
Nutritional factors are one of the interacting factors to affect all developmental aspects among Egyptian children since birth. During the first two years of life, Egyptian studies put more emphasis on child nutrition and development with intensive efforts around breastfeeding because of being a critical period of rapid change. During this phase, studies were implemented to prepare children for subsequent developmental competency in their childhood by investigating the risk factors affecting the early cognitive development of Egyptian infants, and monitoring their cognitive performance. Later on in life, more emphasis was put on either studying factors behind malnutrition or providing educational and nutritional interventions to enhance growth and development.

To address the nutritional needs of school-aged children, global efforts have extensively focused on school-based fortification approaches for school feeding programs (SFPs). SFPs are linked to Goal number 2 (zero hunger) of the Sustainable Development Goals (SDG). The Ministry of Agriculture and Land Reclamation (MOLAR) in Egypt has directed SFP since 1998 to attract children in Egyptian rural areas to attend primary schools by providing them nutritious subsidized in-school meals as a contribution to breakfast consumption. The potential impact goal of targeting children through Food for Education programs (FFE) is to increase their educational achievement and subsequently improve their potential future efficiency and profit. This program includes governmental primary schools within all governorates of Egypt. The close link between nutritional deficiency and diminished cognitive performance and subsequently retarded educational accomplishment was the reason behind implementing nutritional feeding for Egyptian school-aged children to improve their health, cognitive performance, attention span, school attendance, and educational achievement.

Investments in nutrition and cognitive stimulation programs are thus the keys to optimizing child cognitive development and performance. From this perspective, our idea was generated - Relying on the consumption of biscuits that are based on natural ingredients (chickpeas &, peanuts- for improving the cognitive function of children during the school days is much better than relying on drugs.

Both chickpeas and peanuts are types of legumes that are common in Egypt and the middle east. Egypt is a common source for chickpea production in the world where it is mostly consumed as whole seeds and several types of traditional food products. Both of them are overlooked as nutritious food although they have many health benefits as the more expensive nuts and must not be neglected.

These two beans although being nutritionally overachievers that deserve so much more, Yet, they're always moved down to the side-dish zone (e.g puréed of hummus). These two ingredients in addition to Wheat germ and Cinnamon could boost mental health improve mood, memory, cognitive stimulation, muscle control, and other nervous system and brain activities due to their vitamins, minerals, and chemical contents.

The objectives of the study:

to produce a fortified biscuit with chickpea and crushed peanut. To evaluate its effectiveness in terms of its acceptability and impact on cognitive performance for a sample of children aged 8-12 years attending rural primary schools in an Egyptian village after four months of daily intake of 3 biscuits per day for 4 months.

Specific aims To produce Chickpeas and Crushed peanut fortified biscuit To evaluate biscuit effect on short-term and working memory To evaluate biscuit effect on visual memory and the ability for categorization To evaluate biscuit effect on learning for speed of information processing, To evaluate biscuit effect on auditory attention ability with rising levels of difficulty.

Methodology:

Study design and Setting:

The study was a pilot community-based intervention that was conducted in El Othmanyia village of El Mahala district- Gharbyia governorate.

Phases of the study and tools:

This study was conducted in three phases that were done in a simultaneous way. The first phase included children recruitment and baseline assessment before intervention:

Assessment tools (Methods):

Anthropometric measurements of weight and height were carried out to exclude mal-nourished children. All measurements were made according to techniques described in the Anthropometric Standardization Reference Manual. Anthropometric measurements were taken during morning hours on empty stomach before having breakfast or a school meal, within a minimum of 8 hours after micturition and defecation, and after the morning exercises of spine stretching. All scores were calculated based on the WHO growth standards with the help of the Anthro-Program of PC.

Growth assessment according to WHO recommendations

1. Weight (in kg): by a Seca Scale Balance
2. Height (in cm): using Stadiometer
3. BMI (weight/Height2 in meter): calculated Dietary assessment: Detailed nutritional and dietary assessment using Diet Quality index assessment questionnaire, Food frequency pattern, and 24 hours questionnaires.

Cognitive performance assessment: Cognitive performance was assessed before and after the intervention by a battery of psychological tests that covered verbal & non-verbal intelligence, memory, learning, and attention. The children were individually tested by trained researchers.

These tests are:

1. The Digit Span Test: The effect of the intake of the fortified biscuits with stimulation on short-term and working memory was tested by using the Digit Span Test: It is a subtest of the Revised Wechsler Intelligence Scale. The digit span memory task is a verbal measure of immediate memory and working memory maintenance and manipulation. Methodologically, digit span tasks have been proven to be both reliable and valid measures of working memory capacity. The Arabic version of the Revised Wechsler Intelligence Scale for children was used
2. Coding test: It is also a subtest of the Revised Wechsler Intelligence Scale for children. The children had to substitute symbols for numbers as quickly as possible. The score represents the total number of correct symbols written during a fixed time.
3. The auditory vigilance test: which measures the attention ability. It is a measure of the efficiency of identifying signal stimuli in the context of non-signal stimuli. The subjects were asked to pay attention while listening to many words from different categories like a key, ball, school, etc., and they were asked to give a sign, like raising their hands, when they hear certain words, chosen by the administrator. The scores of the test were calculated as total right and totally wrong.
4. The figural memory test: is a measure of free recall of visual objects. The subjects were shown a group of different photos like animals, cars, plants, etc., and they were asked to mention as many photos as they can.

Intervention phase 80 children of those who fulfilled the inclusion and the exclusion criteria were allocated randomly to either one of two groups (every 40 children),

1. The chickpea and crushed peanut biscuits dependent group received one daily pack of three fortified biscuits as snakes between breakfast and lunch on daily basis for four months.
2. The chickpea and crushed peanut biscuits non-dependent group received nothing
3. This supplement was accompanied by cognitive stimulation for both the two groups for the children and their parents (a monthly session with a total of 4 sessions for each)

Composition of the fortified biscuits:

The chickpeas and crushed peanuts fortified biscuit consisted of wheat flour (extract 72%), Chickpeas flour, crushed peanuts, wheat germ, Skimmed milk, corn oil, egg, sugar, Cinnamon, baking powder, salt, and vanilla. The first four constituents help in enhancing immunity, fighting viruses, maintaining regular and healthy bowel movement, regulating blood sugar and cholesterol levels, and more importantly improving the cognitive abilities of school-aged children.

Topics of stimulation sessions I. Sessions for mothers • Sessions for students

• 3. Post Intervention Evaluation Phase This phase included evaluation of the effect of consumption of the chickpea and crushed peanut biscuits on the improvement of the cognitive abilities

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy prepubescent boys and girls in the primary schools with four grades.
* Children should not skip breakfast,
* the number of daily meals (at least 3 times per day),
* does not eat any school snack meal during the school day (other than the biscuits under the study for the fortified biscuits dependent group).

Exclusion Criteria:

* any mental disorder,
* chronic disease,
* visual or auditory impairment, Any malnourished child as detected by both the anthropometric measures and by the Nutritional Status Assessment questionnaire

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Production of Chickpeas and Crushed peanut fortified biscuit | three months after the initiation of the study
  number of fortified biscuits that are based on chickpeas and crushed peanut produced to cover the sampled children on the base of 3 biscuits per day for 4 months to be given to the children to stimulate their cognitive abilities
Mean change of scaled score of the Digit Span Test as a measure of short-term and working memory to detect the fortified biscuits' effect compared to the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase in the mean scaled score of the Digit Span Test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on short-term and working memory. The unpaired t-test between the two means will be used to detect the differences between biscuits dependent and the non-dependent groups.
Mean change of scaled score of the figural memory test as a measure of visual memory to detect the fortified biscuits' effect compared to the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An Increase in the mean scaled score of the figural memory test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on visual memory. The unpaired t-test between the two means will be used to detect the differences between biscuits dependent and the non-dependent groups.
Mean change of scaled score of auditory vigilance tests A and B Test as a measure of auditory attention ability with rising levels of difficulty to detect the fortified biscuits' effect compared to the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase of the mean score of right responses and decrease of the mean score of wrong responses of Auditory vigilance tests A and B Test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on auditory attention. The unpaired t-test between the two means will be to detect the differences between biscuits dependent and the non-dependent groups
Mean change of scaled score of the Coding test as a measure of improved visual-motor coordination, visual encoding, and speed of information processing to detect the fortified biscuits' effect compared to the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase of the mean scaled score of the Coding test indicates an improvement of visual-motor coordination, visual encoding, and speed of information processing as a result of the intake of the fortified biscuits with the cognitive stimulation. The unpaired t-test between the two means will be to detect the differences between biscuits dependent and the non-dependent groups
Mean change of scaled score of the Digit Span Test as a measure of short-term and working memory to detect the fortified biscuits' effect compared to before fortification | 4 months after the initiation of the intervention
  An increase in the mean scaled score of the Digit Span Test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on short-term and working memory. The paired t-test was used to detect the differences between (before and after the intervention)
Mean change of scaled score of the figural memory test as a measure of visual memory to detect the fortified biscuits' effect compared to before fortification | 4 months after the initiation of the intervention
  An Increase in the mean scaled score of the figural memory test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on visual memory. The paired t-test was used to detect the differences between (before and after the intervention)
Mean change of scaled score of auditory vigilance tests A and B Test as a measure of auditory attention ability with rising levels of difficulty to detect the fortified biscuits' effect compared to before fortification | 4 months after the initiation of the intervention
  An increase in the mean score of right responses and decrease in the mean score of wrong responses of Auditory vigilance tests A and B Test as a result of the intake of the fortified biscuits with the cognitive stimulation indicated a positive effect on auditory attention The paired t-test was used to detect the differences between (before and after the intervention)
Mean change of scaled score of the Coding test as a measure of improved visual-motor coordination, visual encoding, and speed of information processing to detect the fortified biscuits' effect compared to before fortification | 4 months after the initiation of the intervention
  An increase in the mean scaled score of the Coding test indicates an improvement of visual-motor coordination, visual encoding, and speed of information processing as a result of the intake of the fortified biscuits with the cognitive stimulation. The paired t-test was used to detect the differences between (before and after the intervention)

SECONDARY OUTCOMES:
Mean change of scaled score of the Digit Span Test as a measure of short-term and working memory to detect the cognitive stimulation effect among the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase in the mean scaled score of the Digit Span Test as a result of cognitive stimulation only indicated a positive effect on short-term and working memory. The paired t-test was used to detect the differences between (before and after the intervention)
Mean change of scaled score of the figural memory test as a measure of visual memory to detect the cognitive stimulation effect among the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An Increase in the mean scaled score of the figural memory test as a result of cognitive stimulation only indicated a positive effect on visual memory. The paired t-test was used to detect the differences between (before and after the intervention)
Change of mean scaled score of Cognitive stimulation ability to improve auditory attention ability with rising levels of difficulty to detect the cognitive stimulation effect among the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase in the mean score of right responses and decrease in the mean score of wrong responses of Auditory vigilance tests A and B Test as a result of cognitive stimulation only indicated a positive effect on auditory attention The paired t-test was used to detect the differences between (before and after the intervention)
Change of mean scaled score of Cognitive stimulation ability to improve learning for speed of information processing to detect the cognitive stimulation effect among the fortified biscuits non-dependent group | 4 months after the initiation of the intervention
  An increase in the mean scaled score of the Coding test indicates an improvement of visual-motor coordination, visual encoding, and speed of information processing as a result of cognitive stimulation only. The paired t-test was used to detect the differences between (before and after the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Ammal M Metwally, PhD (MD), Principal Investigator — National Research Centre of Egypt
Locations (1):
- National Research Centre, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the application for patency
Access Criteria: The data will be accessed through a drive with a link

REFERENCES:
- [Background] El-Din EMS, Elabd MA, Nassar MS, Metwally AM, Abdellatif GA, Rabah TM, Shalaan A, Shaaban SY, Kandeel W, Etreby LAE, Al-Tohamy M. The Interaction of Social, Physical and Nutritive Factors in Triggering Early Developmental Language Delay in a Sample of Egyptian Children. Open Access Maced J Med Sci. 2019 Sep 12;7(17):2767-2774. doi: 10.3889/oamjms.2019.642. eCollection 2019 Sep 15. PMID 31844434
- [Background] Kandeel WA, Rabah TM, Zeid DA, El-Din EMS, Metwally AM, Shaalan A, El Etreby LA, Shaaban SY. Determinants of Exclusive Breastfeeding in a Sample of Egyptian Infants. Open Access Maced J Med Sci. 2018 Oct 2;6(10):1818-1823. doi: 10.3889/oamjms.2018.359. eCollection 2018 Oct 25. PMID 30455755
- [Background] El Din EMS, Rabah TM, Metwally AM, Nassar MS, Elabd MA, Shalaan A, Kandeel W, El Etreby LA, Shaaban SY. Potential Risk Factors of Developmental Cognitive Delay in the First Two Years of Life. Open Access Maced J Med Sci. 2019 Jun 30;7(12):2024-2030. doi: 10.3889/oamjms.2019.566. eCollection 2019 Jun 30. PMID 31406549
- [Background] Metwally AM, Salah El-Din EM, Shehata MA, Shaalan A, El Etreby LA, Kandeel WA, Shaaban SY, Rabah TM. Early Life Predictors of Socio-Emotional Development in a Sample of Egyptian Infants. PLoS One. 2016 Jul 5;11(7):e0158086. doi: 10.1371/journal.pone.0158086. eCollection 2016. PMID 27379907
- [Background] Salah El-Din EM, Monir ZM, Shehata MA, Abouelnaga MW, Abushady MM, Youssef MM, Megahed HS, Salem SME, Metwally AM. A comparison of the performance of normal middle social class Egyptian infants and toddlers with the reference norms of the Bayley Scales -third edition (Bayley III): A pilot study. PLoS One. 2021 Dec 2;16(12):e0260138. doi: 10.1371/journal.pone.0260138. eCollection 2021. PMID 34855785
- [Background] Metwally AM, Shaaban FA, Mahmoud WS, Salah EM, El-Sonbaty MM, Hussien HA, Hamid NA, El Etreby LA, Hassanin A, Monir Z. Vulnerability and Weaknesses of Eating Habits of Overweight School Children as an Entry Risk for COVID-19. Open Access Maced J Med Sci [Internet]. 2020Aug.30 [cited 2020Oct.18];8(T1):158-66. DOI: https://doi.org/10.3889/oamjms.2020.5049 Available from: https://www.id-press.eu/mjms/article/view/5049
- [Background] Metwally AM, El-Sonbaty M, El Etreby LA, El-Din EMS, Hamid NA, Hussien HA, Hassanin A, Monir ZM. Stunting and its Determinants among Governmental Primary School Children in Egypt: A School-based Cross-sectional Study. Open Access Maced J Med Sci [Internet]. 2020 Sep.15 ;8(B):650-7. DOI: https://doi.org/10.3889/oamjms.2020.4757
- [Background] Metwally AM, El-Sonbaty MM, El Etreby LA, Salah El-Din EM, Abdel Hamid N, Hussien HA, Hassanin AM, Monir ZM. Impact of National Egyptian school feeding program on growth, development, and school achievement of school children. World J Pediatr. 2020 Aug;16(4):393-400. doi: 10.1007/s12519-020-00342-8. Epub 2020 Feb 13. PMID 32056148
- [Background] Salah EM, Khalifa AG, Metwally AM, Abdel Hamid N, Hussien HA and Moneer ZM: "The Impact Of School Snacks On Cognitive Function Of Primary School Children In Egypt" Journal of Applied Sciences Research, 8(12): 5639-5650, 2012, ISSN 1819-544X
- [Background] Bundy D, Burbano C, Grosh M, Gelli A, Jukes M, Drake L. Rethinking school feeding: social safety nets, child development, and the education sector. Washington, D.C. (US): The World Food Programme and the World Bank. 2009.
- [Background] WFP (World Food Programme). How school meals contribute to the sustainable development goals. 2017. https://documents.wfp.org/stellent/groups/public/documents/communications/wfp290718.pdf. Accessed 29 Aug 2019.
- [Background] Chavan JK, Kadam SS, Salunkhe DK. Biochemistry and technology of chickpea (Cicer arietinum L.) seeds. Crit Rev Food Sci Nutr. 1986;25(2):107-58. doi: 10.1080/10408398709527449. PMID 3549160
- [Background] Marinangeli CPF, Curran J, Barr SI, Slavin J, Puri S, Swaminathan S, Tapsell L, Patterson CA. Enhancing nutrition with pulses: defining a recommended serving size for adults. Nutr Rev. 2017 Dec 1;75(12):990-1006. doi: 10.1093/nutrit/nux058. PMID 29202192
- [Background] Arya SS, Salve AR, Chauhan S. Peanuts as functional food: a review. J Food Sci Technol. 2016 Jan;53(1):31-41. doi: 10.1007/s13197-015-2007-9. Epub 2015 Sep 19. PMID 26787930
- [Background] Moreira-Rosario A, Pinheiro H, Calhau C, Azevedo LF. Can wheat germ have a beneficial effect on human health? A study protocol for a randomised crossover controlled trial to evaluate its health effects. BMJ Open. 2016 Nov 10;6(11):e013098. doi: 10.1136/bmjopen-2016-013098. PMID 28157671
- [Background] Rao PV, Gan SH. Cinnamon: a multifaceted medicinal plant. Evid Based Complement Alternat Med. 2014;2014:642942. doi: 10.1155/2014/642942. Epub 2014 Apr 10. PMID 24817901
- [Background] Lee EJ, Chen HY, Hung YC, Chen TY, Lee MY, Yu SC, Chen YH, Chuang IC, Wu TS. Therapeutic window for cinnamophilin following oxygen-glucose deprivation and transient focal cerebral ischemia. Exp Neurol. 2009 May;217(1):74-83. doi: 10.1016/j.expneurol.2009.01.019. Epub 2009 Feb 5. PMID 19416670
- [Background] Lohman, T.G., A.F. Roche, R. Martorell. Anthropometric standardization reference manual.Champaign, IL: Human kinetics Publishers. 1988.
- [Background] Pollitt, E., Methods for the behavioral assessment of the consequences of malnutrition. In Lockwood ER & Scrimshaw NS (eds): Methods of the evaluation of the impact of food and nutrition programs. Tokyo, UNU. 1984
- [Background] Newby PK, Hu FB, Rimm EB, Smith-Warner SA, Feskanich D, Sampson L, Willett WC. Reproducibility and validity of the Diet Quality Index Revised as assessed by use of a food-frequency questionnaire. Am J Clin Nutr. 2003 Nov;78(5):941-9. doi: 10.1093/ajcn/78.5.941. PMID 14594780
- [Background] Wechsler, D.,. Manual for the Wechsler Intelligence Scale for Children - Revised (WISC-R), the Psychological Corporation, NY. 1977.
- [Background] Cserjesi R, Molnar D, Luminet O, Lenard L. Is there any relationship between obesity and mental flexibility in children? Appetite. 2007 Nov;49(3):675-8. doi: 10.1016/j.appet.2007.04.001. Epub 2007 Apr 10. PMID 17543417
- [Background] Ahmed HH, Abla G. Khalifa AG, Eskander EF, Sayed AH and Abdel-Nabi IM. Biochemical and neurological effects of obesity on primary school girls. Nature and Science 2010;8(4)
- [Background] Babikian T, Boone KB, Lu P, Arnold G. Sensitivity and specificity of various digit span scores in the detection of suspect effort. Clin Neuropsychol. 2006 Feb;20(1):145-59. doi: 10.1080/13854040590947362. PMID 16393925
- [Background] de Paula JJ, Malloy-Diniz LF, Romano-Silva MA. Reliability of working memory assessment in neurocognitive disorders: a study of the Digit Span and Corsi Block-Tapping tasks. Braz J Psychiatry. 2016 Jul-Sep;38(3):262-3. doi: 10.1590/1516-4446-2015-1879. No abstract available. PMID 27579598
- [Background] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997
- [Background] Ismaiel, E and M. Kamel. Wechsler Intelligence Scale for Children Revised, Arabic version. El-Nahda El massryia, Cairo; 1993.
- [Background] Sattler, J.M. Assessment of children: Revised and updated (3rd ed.). San Diego: Jerome M. Sattler, Publisher, Inc. 1992
- [Background] Yunis, F.A., A.G. Khalifa, Z.M. Monir, A.A. Ayad, S.A. Gabr. Physical growth, nutritional status and intellectual performance among school children of a rural village. Med J Cairo Univ., 1995; 63(4): 971-80.
- [Background] Wahba, S.A. and A.G. Khalifa. Breakfast skipping and cognitive functions of primary school children, relation to nutritional status. The Gaz Egypt Paed, 1998; 46(3,4): 203-16
- [Background] Khalifa, A.G., F. Hasaballa, S. Tawfik and M. Mansour. Nutritional Status and Cognitive Performance of Primary School Children, Relationship to Social Status and Academic Achievement. JAC, 2001; 12(1): 31-54
- [Background] Samer M. Al-Zoubi, Mohammad A. Bani Younes (2015). Low Academic Achievement: Causes and Results. Theory and Practice in Language Studies, Vol. 5, No. 11, pp. 2262-2268
- [Background] Puerta, L. (2015). Relationship between cognitive processes and academic performance in high school students. Psychologia: Avances de la Disciplina, 9(2), 85-100
- [Background] MeenuDev. (2016) Factors Affecting the Academic Achievement: A Study of Elementary School Students of NCR Delhi, India. Journal of Education and Practice. Vol.7, No.4, pp. 70-74
- [Background] Frolek Clark, G. G., Schlabach, T. L., Barnett, M. E., Carr, M. A., Hinkle, B. L., Kluever, J. L., … Kluever, A. L. (2011, August). American Occupational Therapy Association, Inc. Retrieved from www.aota.org
- See also: https://documents.wfp.org/stellent/groups/public/documents/communications/wfp290718.pdf. — https://documents.wfp.org/stellent/groups/public/documents/communications/wfp290718.pdf.
- See also: WHO, AnthroPlus for personal computers. Manual Software for assessing growth of the world's children and adolescents 2009. Geneva — http://www.who.int/growthref/tools/en/